CLINICAL TRIAL: NCT05379998
Title: Comparison of Neural Mobilization and Proprioceptive Neuromuscular Facilitation Hold Relax Technique on Lower Limb Motor Function in Hemiplegic Stroke
Brief Title: Neural Mobilization Versus PNF Hold Relax Technique on Lower Extremity in Hemiplegic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01244 Nida khan
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Hemiplegic Stroke
Keywords: Neural mobilization; PNF hold relax; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: This will be a single blinded study. The data will be coded and the analyst will also be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A(neural mobilization) (Experimental): sciatic nerve mobilization(sliding technique)
  Interventions: Other: Neural mobilization
- Group B(PNF hold relax) (Experimental): PNF hold relax technique of Hamstring muscle
  Interventions: Other: PNF hold relax technique

INTERVENTIONS:
Other: Neural mobilization — Sciatic nerve mobilization (sliding technique) will be performed by a physical therapist. The sciatic nerve mobilization technique improves the nerve mobility of the hemiparetic lower limb in a nervous system patient and is helpful in increasing the ROM of the lower limbs without resistance.
  Arms: Group A(neural mobilization)
Other: PNF hold relax technique — Proprioceptive neuromuscular facilitation hold relaxation technique of hamstring muscle will be performed by the physical therapist three days a week for 6 weeks. In the hold relax technique after reaching the point of resistance, an isometric contraction is performed against the resistance to get a pain free response.
  Arms: Group B(PNF hold relax)

SUMMARY:
Several studies about the effects of nerve mobilizations and stretching exercises have been conducted. This study will contribute to describing the long term effects of these techniques on gait, motor function and quality of life in hemiplegic stroke patients and compare the effectiveness of both techniques.

DETAILED DESCRIPTION:
Several studies about the effects of nerve mobilizations and stretching exercises have been conducted. Evidence regarding the comparison of these two techniques is sparse and is based on different clinical experiences and a less number of studies with limited methodological design. There has been no work regarding the long term effects of these two techniques in improving lower limb motor function in Hemiplegic stroke patients. This study will contribute to describing the long term effects of these techniques on gait, motor function and quality of life in hemiplegic stroke patients and compare the effectiveness of both techniques. A total of 54 patients diagnosed with Hemiplegic stroke will be selected for the collection of data according to the inclusion criteria. Patients will be divided into two groups, Group A and Group B. Group A will receive sciatic nerve mobilization (sliding technique) and Group B will receive Proprioceptive neuromuscular mobilization Hold relax technique 3 days a week for 30 mins per day for 6 weeks. Sciatic nerve mobilizations (sliding technique) will be performed for a duration of 1 minute each for 6 such sets with 60 seconds rest period followed by every set. The Hold Relax Technique of Hamstring will be performed with each hold period lasting for 10 seconds followed by a relaxation phase of 10-15 seconds for 10 repetitions. Data will be collected at baseline, after 3weeks and at 6 weeks after intervention from both groups. Gait will be measured using TUG (Timed up and go), Quality of life will be measured using the Urdu version of SS-QOL(stroke-specific quality of life)and lower limb motor function will be measured using fugl Meyer scale(lower extremity)

ELIGIBILITY:
Inclusion Criteria:

* Patients with subacute to chronic (3-12months) Hemiplegic Stroke.
* Both Genders.
* Age between 20 and 70 years.
* Patients classified as grade 2 and 3 as per the Modified Rankin scale.
* Patients with or without assistive devices.

Exclusion Criteria:

* Patients having cardiac disorders, rheumatic and orthopedic diseases that would impede the performance of the technique.
* Patients who have undergone some surgery recently.
* Patients having cognitive impairments.
* Contractures of the lower limb joints.
* Patients having associated Neurological Pathologies.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Fugl meyer(lower extremity) | baseline
  The Fugl-Meyer Assessment is the most widely used standardized clinical scale designed to assess motor function, balance, sensation qualities and joint function in hemiplegic post-stroke patients. The total motor score ranges from 0 to 100 including 28 points for the lower extremity and 6 scores for coordination/speed. Sensation score ranges from 0 to 12, joint range of motion from 0 to 20 and joint pain from 0 to 20.
Fugl meyer(lower extremity) | 3 weeks
  The Fugl-Meyer Assessment is the most widely used standardized clinical scale designed to assess motor function, balance, sensation qualities and joint function in hemiplegic post-stroke patients. The total motor score ranges from 0 to 100 including 28 points for the lower extremity and 6 scores for coordination/speed. Sensation score ranges from 0 to 12, joint range of motion from 0 to 20 and joint pain from 0 to 20.
Fugl meyer(lower extremity) | 6 weeks
  The Fugl-Meyer Assessment is the most widely used standardized clinical scale designed to assess motor function, balance, sensation qualities and joint function in hemiplegic post-stroke patients. The total motor score ranges from 0 to 100 including 28 points for the lower extremity and 6 scores for coordination/speed. Sensation score ranges from 0 to 12, joint range of motion from 0 to 20 and joint pain from 0 to 20.
Timed up and go (TUG) | baseline
  The timed up and Go test (TUG) is a sensitive and specific measure of the probability of falls among older adults. This test is simple and used to measure the risk of falls, and the progress of walking, balance and sit to stand. The TUG is a reliable, valid, and easy-to-administer clinical tool for assessing advanced functional mobility after a stroke.<10sec shows complete independence for ambulation and transfers (with and without walking aid). An older adult who takes ≥12 seconds to complete the TUG is at risk of falling.
Timed up and go (TUG) | 3 weeks
  The timed up and Go test (TUG) is a sensitive and specific measure of the probability of falls among older adults. This test is simple and used to measure the risk of falls, and the progress of walking, balance and sitting to stand. The TUG is a reliable, valid, and easy-to-administer clinical tool for assessing advanced functional mobility after a stroke.<10sec shows complete independence for ambulation and transfers (with and without walking aid). An older adult who takes ≥12 seconds to complete the TUG is at risk of falling.
Timed up and go (TUG) | 6 weeks
  The timed up and Go test (TUG) is a sensitive and specific measure of the probability of falls among older adults. This test is simple and used to measure the risk of falls, and the progress of walking, balance and sitting to stand. The TUG is a reliable, valid, and easy-to-administer clinical tool for assessing advanced functional mobility after a stroke.<10sec shows complete independence for ambulation and transfers (with and without walking aid). An older adult who takes ≥12 seconds to complete the TUG is at risk of falling.
Stroke specific quality of life (SS-QOL) | baseline
  Stroke specific quality of life (SS-QOL) is a standard scale used to evaluate health as related to the quality of life, particularly in stroke patients. Urdu version of the stroke-specific quality of life scale will be used. The total score ranges from 49 to 245 with higher scores indicating higher quality of life. The minimum score is 49.
Stroke specific quality of life (SS-QOL) | 3 weeks
  Stroke specific quality of life (SS-QOL) is a standard scale used to evaluate health as related to the quality of life, particularly in stroke patients. Urdu version of the stroke-specific quality of life scale will be used. The total score ranges from 49 to 245 with higher scores indicating higher quality of life. The minimum score is 49.
Stroke specific quality of life (SS-QOL) | 6 weeks
  Stroke specific quality of life (SS-QOL) is a standard scale used to evaluate health as related to the quality of life, particularly in stroke patients. Urdu version of the stroke-specific quality of life scale will be used. The total score ranges from 49 to 245 with higher scores indicating higher quality of life. The minimum score is 49.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Holly Family Hospital, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No